CLINICAL TRIAL: NCT02368795
Title: Non-inferiority Trial Comparing Pharmacological Prevention Alone Versus Pancreatic Stents Plus Pharmacological Prevention to Prevent Post-ERCP Pancreatitis
Brief Title: Non-inferiority of Pharmacological Prevention Alone Versus Pancreatic Stents to Prevent Post-ERCP Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 642416
Record Dates: First submitted 2015-02-02; First posted 2015-02-23 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Pancreatitis
Keywords: Endoscopic Retrograde Cholangiopancreatography; Pancreatic duct stenting; Post-ERCP pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Indomethacin; Isosorbide Dinitrate; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacological Prevention (Placebo Comparator): Combination of rectal indomethacin, sublingual isosorbide dinitrate and intravenous hydration with Ringer's lactate serum without pancreatic stenting
  Interventions: Drug: Indomethacin; Drug: Isosorbide Dinitrate; Drug: Ringer's lactate
- Pancreatic Stent (Active Comparator): Pancreatic Stent PLUS Pharmacological Prevention
  Interventions: Device: Pancreatic Stent; Drug: Indomethacin; Drug: Isosorbide Dinitrate; Drug: Ringer's lactate

INTERVENTIONS:
Device: Pancreatic Stent — A 5-Fr, 4-cm-long stent (Endoflex) with a single duodenal pigtail is used for pancreatic duct stenting
  Arms: Pancreatic Stent
Drug: Indomethacin — Indomethacin 100 mg suppository ten minutes before ERCP
Drug: Isosorbide Dinitrate — Sublingual Isosorbide dinitrate 5 mg before ERCP
Drug: Ringer's lactate — IV Ringer's lactate serum with a dose of 6 cc/kg/h during the procedure and 20 cc/kg after ERCP as a bolus dose and 3 cc/kg/h for the next 8 hours.

SUMMARY:
Pancreatitis is the most important complication of ERCP. The severity of this condition varies from mild to severe and can lead to prolonged hospitalization, surgical interventions, and even death. Several patient-related and procedure related factors have been identified that are associated with a higher risk of post-ERCP pancreatitis. So far, several methods have been proposed to avoid pancreatitis in patients at higher risk of this complication.

Several studies have shown that different drug therapies (indomethacin suppository, a sublingual nitrate tablet and the administration of intravenous Ringer's solution) each may reduce the incidence of post-ERCP pancreatitis. All these drug therapies are safe, cheap and easy to administer.

Several other studies have shown that pancreatic duct stenting (placement of a plastic tube in the pancreatic duct) is an effective intervention in preventing and reducing the severity of post-ERCP pancreatitis, especially in high-risk groups. However, there are still a few drawbacks to consider with pancreatic duct stenting: there are some difficulties with insertion of a PD stent, it is associated with a need for radiological follow-up and/or repeat endoscopy for removal, higher cost and a small but important risk of complications (e.g. stent migration).

Most of the clinical trials of pancreatic duct stenting were performed, before the results of trials of drug therapies were available. Moreover, no RCT (to the investigators knowledge) has compared the efficacy of pancreatic duct stenting in patients who already received a combination of drug therapies to prevent post-ERCP pancreatitis in high-risk patients. The purpose of this study is to determine the noninferiority of a combination of drug therapies in relation to pancreatic duct stenting to prevent post-ERCP pancreatitis in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

Patients at high risk of post-ERCP Pancreatitis undergoing ERCP are eligible to enter the study. At least one major or two minor criteria must be present for the patient to be considered at high risk for PEP:

Major

* Sphincter of Oddi dysfunction.
* History of previous PEP.
* Pancreatic injection.
* Precut sphincterotomy.
* Balloon sphincter dilation without sphincterotomy.
* Pancreatic guidewire passages > 1.

Minor

* Female patients aged<60 years.
* Nondilated common bile duct (CBD).
* Normal serum bilirubin (<2mg/dl).
* Failure to clear bile duct stones.
* Failed cannulation.
* Difficult cannulation (Time to CBD cannulation more than 10 min or more than five attempts at cannulation).

Exclusion Criteria:

* Age younger than 15 years.
* History of sphincterotomy.
* Surgically altered anatomy (Billroth II gastrectomy or Roux-en-Y anastomosis).
* Uncontrolled coagulopathy.
* Tumor of ampulla of Vater.
* Those undergoing routine biliary-stent exchange.
* Acute pancreatitis at the time of ERCP.
* Chronic pancreatitis.
* Regular NSAID use during preceding week.
* Unable to tolerate indomethacin (Creatinine level >1.4 mg/dL or active peptic ulcer disease).
* Unable to tolerate nitrates (closed-angle glaucoma).
* Unable to tolerate aggressive hydration (cardiac insufficiency: NYHA FC II or higher, renal insufficiency, electrolyte disturbances, clinical signs of fluid overload including peripheral or pulmonary edema, liver dysfunction with varix>F1, or respiratory insufficiency).
* Patients requiring pancreatic duct drainage: to bridge dominant strictures, bypass obstructing pancreatic duct stones, drain pseudocysts, seal duct disruptions, pancreatic head cancer with main PD obstruction, IPMN or Pancreas divisum.
* Known main pancreatic duct stricture toward the head of pancreas.
* Pregnancy or breastfeeding.
* Refusal to participate in the study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Post-ERCP pancreatitis | 24 hours after ERCP
  Pancreatitis is defined as new or worsened abdominal pain and tenderness with amylase levels at least three times above the upper limit of normal at 24 hours after the procedure, requiring hospital admission or a prolongation of planned admission.

SECONDARY OUTCOMES:
Severity of acute pancreatitis according to revised Atlanta classification (Banks et al. GUT 2013) | One week after ERCP
  Mild acute pancreatitis (No organ failure, No local or systemic complications) Moderately severe acute pancreatitis (transient organ failure that resolves within 48 h and/or Local or systemic complications without persistent organ failure) Severe acute pancreatitis (Persistent organ failure >48 h)

CONTACTS AND LOCATIONS:
Locations (1):
- Shariati hospital, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Sotoudehmanesh R, Ali-Asgari A, Khatibian M, Mohamadnejad M, Merat S, Sadeghi A, Keshtkar A, Bagheri M, Delavari A, Amani M, Vahedi H, Nasseri-Moghaddam S, Sima A, Eloubeidi MA, Malekzadeh R. Pharmacological prophylaxis versus pancreatic duct stenting plus pharmacological prophylaxis for prevention of post-ERCP pancreatitis in high risk patients: a randomized trial. Endoscopy. 2019 Oct;51(10):915-921. doi: 10.1055/a-0977-3119. Epub 2019 Aug 27. PMID 31454851